CLINICAL TRIAL: NCT03101566
Title: A Multi-Center Randomized Phase II Study of Nivolumab in Combination With Gemcitabine/Cisplatin or Ipilimumab as First Line Therapy for Patients With Advanced Unresectable Biliary Tract Cancer [CA209-9FC]
Brief Title: Study of Nivolumab in Combination With Gemcitabine/Cisplatin or Ipilimumab for Patients With Advanced Unresectable Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.026; HUM00126271 (Other: University of Michigan); HUM00130035 (Other: University of Michigan)
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-09

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gemcitabine + Cisplatin + Nivolumab (Experimental): Drug: Gemcitabine 1000 mg/m2 IV on days 1,8 every 3 weeks
  Drug: Cisplatin 25 mg/m2 IV on days 1,8 every 3 weeks
  Drug: Nivolumab 360 mg IV on day 1 every 3 weeks
  If there is continued benefit after 6 months, then:
  Drug: Nivolumab 240 mg IV on day 1 every 2 weeks
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Nivolumab
- Nivolumab + Ipilimumab (Experimental): Drug: Ipilimumab
  1 mg/kg IV on day 1 every 6 weeks
  Drug: Nivolumab 240 mg IV on day 1 every 2 weeks
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 IV
  Arms: Gemcitabine + Cisplatin + Nivolumab
Drug: Cisplatin — Cisplatin 25 mg/m2 IV
  Arms: Gemcitabine + Cisplatin + Nivolumab
Drug: Ipilimumab — Ipilimumab 1 mg/kg IV
  Arms: Nivolumab + Ipilimumab
Drug: Nivolumab — Nivolumab 360 mg or 240 mg IV

SUMMARY:
The purpose of this trial is to evaluate the effect of investigational drug nivolumab in combination with either gemcitabine/cisplatin chemotherapy, or in combination with another investigational agent ipilimumab in patients with advanced unresectable biliary tract cancer.

Gemcitabine/cisplatin is the standard of care treatment for biliary tract cancer.

Nivolumab and ipilimumab are types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack the cancer cells. Nivolumab (Opdivo) is FDA approved for the treatment of several cancers including metastatic melanoma, advanced lung, kidney, head & neck and bladder cancer. The combination of nivolumab and ipilimumab (Yervoy) is FDA approved for metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically confirmed adenocarcinoma of the biliary tract (intra-hepatic, extra-hepatic (hilar, distal) or gall bladder) that is not eligible for curative resection, transplantation, or ablative therapies. Tumors of mixed histology are excluded.
* Patients may have received prior radiation, chemoembolization, radioembolization or other local ablative therapies or hepatic resection if completed ≥ 4 weeks prior to registration AND if patient has recovered to <= grade 1 toxicity. Extrahepatic palliative radiation is permitted if completed ≥ 2 weeks prior to enrollment AND if patient has recovered to ≤ grade 1 toxicity.
* Patients must have radiographically measurable disease in at least one site not previously treated with radiation or liver directed therapy (including bland, chemo- or radio-embolization, or ablation) either within the liver or in a metastatic site.
* Must be ≥18 years of age
* Must have a Child-Pugh score of A (prognosis in chronic liver disease and cirrhosis)
* Must have an ECOG (Eastern Cooperative Oncology Group) performance status of 0-1
* Ability to understand and willingness to sign IRB-approved informed consent
* Willing to provide archived tissue, if available, from a previous diagnostic biopsy
* Must be able to tolerate CT (computerized tomography) and/or MRI (magnetic resonance imaging) with contrast
* Must have adequate organ function obtained ≤ 2 weeks prior to registration

Exclusion Criteria:

* Patients may not have received prior systemic treatment (chemotherapy or targeted therapy) for advanced BTC (biliary tract cancer). Prior adjuvant chemotherapy is permitted provided it was completed > 6 months from registration.
* Must not have a diagnosis of immunodeficiency, or have received systemic steroid therapy, or any other form of immunosuppressive therapy within 7 days prior to trial treatment.
* Must not have known Hepatitis B, Hepatitis C, or HIV seropositivity. Testing is not required in absence of clinical suspicion.
* Must not have prior history of organ transplantation or brain metastasis.
* Must not have undergone a major surgical procedure < 4 weeks prior to registration.
* Must not have an active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ. Patients with history of malignancy are eligible provided primary treatment of that cancer was completed > 1 year prior to registration and the patient is free of clinical or radiologic evidence of recurrent or progressive malignancy.
* Must have no ongoing active, uncontrolled infections
* Must not have received a live vaccine within 30 days of planned start of the study therapy.
* Must not have a psychiatric illness, other significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements.
* Women must not be pregnant or breastfeeding since study drugs may harm the fetus or child.
* Women of child-bearing potential and men must agree to use 2 methods of adequate contraception (hormonal plus barrier or 2 barrier forms) OR abstinence prior to study entry, for the duration of study participation and for 5 months (for women) and 7 months (for men) following completion of study therapy.
* Participants with an active, known or suspected autoimmune disease which may affect vital organ function, or has/may require systemic immunosuppressive therapy for management are excluded. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 7 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav Sahai, MBBS, MS, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (7):
- United States (7):
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahai V, Griffith KA, Beg MS, Shaib WL, Mahalingam D, Zhen DB, Deming DA, Zalupski MM. A randomized phase 2 trial of nivolumab, gemcitabine, and cisplatin or nivolumab and ipilimumab in previously untreated advanced biliary cancer: BilT-01. Cancer. 2022 Oct 1;128(19):3523-3530. doi: 10.1002/cncr.34394. Epub 2022 Jul 27. PMID 35895381

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine + Cisplatin + Nivolumab: Gemcitabine1000 mg/m2 IV and Cisplatin 25 mg/m2 IV on days 1 and 8 every 3 weeks + Nivolumab 360 mg IV on day 1 every 3 weeks for up to 8, 3-week cycles. Followed by Nivolumab alone at 240 mg IV every 2 weeks. Total duration no longer than 2 years of study treatment.
- Nivolumab + Ipilimumab: Nivolumab 240 mg IV on day 1 every 2 weeks + Ipilimumab 1 mg/kg IV on day 1 every 6 weeks; for up to 2 years in absence of disease progression.
Period: Overall Study
Arm/Group | Gemcitabine + Cisplatin + Nivolumab | Nivolumab + Ipilimumab
Started | 37 | 38
Received at Least One Dose of Protocol Therapy | 35 | 33
Assessed for Primary and Secondary Progression-free Survival | 32 | 33
Completed | 31 | 31
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine + Cisplatin + Nivolumab | Nivolumab + Ipilimumab | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Full Range); unit: years] | 59 [20 to 80] | 61 [34 to 79] | 60 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 20 | 18 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 31 | 36 | 67
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 32 | 28 | 60
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Disease status at enrollment [Count of Participants; unit: Participants]
  locally advanced | 4 | 4 | 8
  metastatic | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Alive and Without Progression at 6 Months Following the Initiation of Treatment
Description: The primary endpoint is PFS (Progression Free Survival) at 6 months following the initiation of treatment. Progression will be defined clinically or on imaging as per immune related response evaluation criteria in solid tumors (irRECIST) definition.
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine + Cisplatin + Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 32 | 33
percentage of participants | 59.4 [40.5 to 74] | 21.2 [9.4 to 36.3]
Statistical Analysis 1: Comparison: Gemcitabine + Cisplatin + Nivolumab vs Nivolumab + Ipilimumab; Test type: Other; PFS at 6 months was estimated for this trial using the product-limit method of Kaplan and Meier with 95% confidence intervals calculated using Greenwood's formula. All statistical analyses were completed using the SAS System, v9.4 [Cary, NC, USA]

2. Secondary Outcome: Median Progression Free Survival Time
Description: The median time patients are alive without progression following the initiation of treatment wherein progression will be defined clinically or on imaging as per irRECIST criteria.
Time Frame: Patients will be followed until death, withdrawal from study, or until 2 years, whichever is earliest
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gemcitabine + Cisplatin + Nivolumab: Drug: Gemcitabine 1000 mg/m2 IV on days 1,8 every 3 weeks
  Drug: Cisplatin 25 mg/m2 IV on days 1,8 every 3 weeks
  Drug: Nivolumab 360 mg IV on day 1 every 3 weeks
  If there is continued benefit after 6 months, then:
  Drug: Nivolumab 240 mg IV on day 1 every 2 weeks
  Gemcitabine: Gemcitabine 1000 mg/m2 IV
  Cisplatin: Cisplatin 25 mg/m2 IV
  Nivolumab: Nivolumab 360 mg or 240 mg IV
- Nivolumab + Ipilimumab: Drug: Ipilimumab
  1 mg/kg IV on day 1 every 6 weeks
  Drug: Nivolumab 240 mg IV on day 1 every 2 weeks
  Ipilimumab: Ipilimumab 1 mg/kg IV
  Nivolumab: Nivolumab 360 mg or 240 mg IV
Arm/Group | Gemcitabine + Cisplatin + Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 35 | 33
months | 6.6 [3.4 to 7.7] | 3.9 [2.3 to 4.5]

3. Secondary Outcome: Median Overall Survival Time
Description: The median overall survival time following the initiation of treatment.
Time Frame: Patients will be followed until death, withdrawal from study, or until 2 years, whichever is earliest
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Cisplatin + Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 32 | 33
months | 10.6 [6.4 to 24.5] | 8.2 [5.8 to 16.9]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate will be determined as per the combined RECIST v1.1 and irRECIST criteria
Time Frame: Up to two years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Gemcitabine + Cisplatin + Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 33 | 32
percentage of patients | 22.9 [10.4 to 40.1] | 3.0 [0.1 to 15.8]

ADVERSE EVENTS:
Time Frame: Data on adverse events was collected from the time of the initial study treatment administration through 100 days after the last dose of study treatment. Any serious adverse event that occured more than 100 days after the last study treatment and is considered related to the study treatment or intervention is also reported.
Arm/Group | Gemcitabine + Cisplatin + Nivolumab | Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 22/35 | 23/33
Serious Adverse Events (participants affected / at risk) | 25/35 | 23/33
Other Adverse Events (participants affected / at risk) | 34/35 | 28/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin + Nivolumab (N=35) | Nivolumab + Ipilimumab (N=33)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 4 (4) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (3) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 3 (4) | 3 (4)
Sepsis (Infections and infestations) | 4 (6) | 2 (3)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (3) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine + Cisplatin + Nivolumab (N=35) | Nivolumab + Ipilimumab (N=33)
Anemia (Blood and lymphatic system disorders) | 16 | 5
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 1 | 3
Papilledema (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 14 | 11
Ascites (Gastrointestinal disorders) | 1 | 5
Bloating (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 13 | 10
Diarrhea (Gastrointestinal disorders) | 13 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 3 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 3
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 18 | 9
Vomiting (Gastrointestinal disorders) | 10 | 5
Chills (General disorders) | 3 | 2
Edema limbs (General disorders) | 8 | 8
Fatigue (General disorders) | 15 | 16
Fever (General disorders) | 7 | 4
Flu like symptoms (General disorders) | 1 | 3
Infusion related reaction (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 4 | 0
Pain (General disorders) | 7 | 5
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 2
Infections and infestations - Other, specify (Infections and infestations) | 4 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 8 | 5
Alkaline phosphatase increased (Investigations) | 7 | 6
Aspartate aminotransferase increased (Investigations) | 5 | 4
Blood bilirubin increased (Investigations) | 2 | 6
Creatinine increased (Investigations) | 3 | 3
Investigations - Other, specify (Investigations) | 0 | 2
Lipase increased (Investigations) | 2 | 1
Lymphocyte count decreased (Investigations) | 4 | 2
Neutrophil count decreased (Investigations) | 14 | 0
Platelet count decreased (Investigations) | 11 | 0
Weight gain (Investigations) | 1 | 2
Weight loss (Investigations) | 7 | 6
White blood cell decreased (Investigations) | 8 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 9
Dehydration (Metabolism and nutrition disorders) | 6 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 9 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 3 | 2
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 2
Anxiety (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 8
Hot flashes (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 5 | 0
Hypotension (Vascular disorders) | 3 | 1
Phlebitis (Vascular disorders) | 2 | 0
Thromboembolic event (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT03101566/Prot_SAP_000.pdf